CLINICAL TRIAL: NCT06638476
Title: Step Training in Persons Post-stroke
Brief Title: Lateral Perturbation Induced Step Training Compared to Lateral Voluntary Step Training in People with Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vicki Gray (Other)
Responsible Party: Sponsor-Investigator, Vicki Gray, Associate Professor, University of Maryland, Baltimore
Organization: University of Maryland, Baltimore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00056550; American Heart Association (Other Grant/Funding Number: 14CRP19880025); H133P100014, H133F140027 (Other Grant/Funding Number: National Institute on Disability, Independent Living and Rehabilitation Research); P30AG028747 (NIH)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: balance; exercise; falls; stroke
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perturbation induced step training (Experimental): Participants will receive 18 sessions over 6 weeks.
  Interventions: Other: Perturbation Induced Step training
- Voluntary Step training (Active Comparator): Participants will receive 18 sessions over 6 weeks.
  Interventions: Other: Voluntary step training

INTERVENTIONS:
Other: Perturbation Induced Step training — A sudden lateral displacement of the treadmill.
  Arms: Perturbation induced step training
Other: Voluntary step training — Voluntary steps emphasizing speed, movement of center of mass and taking larger steps.
  Arms: Voluntary Step training

SUMMARY:
The goal of this clinical trial is to see if perturbation-induced step training improves stepping performance during a reactive and voluntary step. The main questions it aims to answer are:

Does perturbation induced step training improve step initation time and first recovery step?

Researchers will compare lateral perturbation induced step training to lateral voluntary step training to see if the first recovery steps improve.

Participants will:

Vist the lab for an initial assessment, post exercise and one month post exercise of voluntary and perturbation induced stepping performance, and clinical tests of balance, motor recovery, sensory and strength tests.

Exercise 3 times a week for 6 weeks in person

Track falls for 6 months after the exercise.

DETAILED DESCRIPTION:
Stroke is the leading cause of disability in the United States as the result of an increased survival rate over the last 25 years. A high frequency of falls is commonly reported in this group due to the residual sensorimotor deficits and impairments to balance. Many falls occur when weight is transferred laterally and an equal number of falls happen during voluntary movements as during unexpected disturbances such as a trip, push or pull. Typically, either will involve a protective step to recover balance. Thus, the purpose of this study is to compare the effects of reactive lateral step training to voluntary lateral step training on the performance of the protective step, functional balance and falls in persons post-stroke. Thirty participants with a stroke will be randomized to one of two interventions, reactive step training or voluntary step training. In the voluntary step training group, participants will perform voluntary steps. In the reactive step training group, participants will perform reactive steps generated by the Active Step. The training will be 3 times a week for 6 weeks. The step initiation time, will be compared in both the voluntary and reactive steps at baseline before the intervention, post-intervention and a test of retention will occur one month after the training. Functional balance will be assessed with the Community Balance & Mobility Scale and falls will be compared in the 6 months preceding the intervention to 6 months post-intervention testing. If reactive step training is effective, then the protective step characteristics, functional balance and the number of falls will be reduced compared to the voluntary step training group.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis as a result of a stroke greater than 6 months previous to the study
* Able to walk 10 meters with or without a walking aid
* Have the cognitive ability to give informed consent

Exclusion Criteria:

* Medical condition precluding participation in regular exercise, such as acute cardiac or respiratory conditions limiting activity and other health conditions significantly impacting the ability to walk beyond the effects of the stroke, such as other neurological conditions or peripheral neuropathies.
* Bilateral stroke or a previous stroke in the contralateral hemisphere.
* Aphasia

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Step initiation time | Baseline, 6 weeks
  Change in Step initiation time measured from the time of the puller or light cue onset to the first foot off the force platform.
First step length | Baseline, 6 weeks
  Global step length based on the displacement of the ankle marker normalized by the participants height.

SECONDARY OUTCOMES:
step velocity | Baseline, 6 weeks
  The step displacment divided by the time to complete the first step
Step clearance | Baseline, 6 weeks
  The vertical displacment of the ankle marker normalized the the body height.
Community Balance & Mobility Scale | Baseline, 6 weeks
  Balance measure
Activities Specific Balance Confidence | Baseline, 6 weeks
  A self reported measure of balance confidence
Falls | 6 months pre-enrollment, 6 months post exercise
  Number of falls

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore, Baltimore, MD, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The data was collected more than 5 years ago.